CLINICAL TRIAL: NCT01842906
Title: Randomized Controlled Trial for Assessment of a Novel Non-Pharmacologic Intervention for Decrease in Altitude Illness
Brief Title: Study Looking at End Expiratory Pressure for Altitude Illness Decrease (SLEEP-AID)
Acronym: SLEEP-AID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Grant S Lipman, Clinical Associate Professor of Emergency Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SLEEP-AID
Record Dates: First submitted 2013-04-22; First posted 2013-04-30 (Estimated); Results first posted 2017-04-20 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-11

CONDITIONS: Acute Mountain Sickness
Keywords: positive end expiratory pressure; acute mountain sickness; prevention; high altitude
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Theravent (Experimental): A singe use, disposable, positive end expiratory pressure device worn over the nostrils while sleeping.
  Interventions: Device: Theravent
- Control (Sham Comparator): A visibly identical sham device that does not provide positive end expiratory pressure.
  Interventions: Device: Control

INTERVENTIONS:
Device: Theravent — nasal EPAP device
  Arms: Theravent
Device: Control — Sham device without EPAP
  Arms: Control

SUMMARY:
The study is examining if an over-the-counter device (Theravent) worn while sleeping can reduce acute mountain sickness upon awakening in a high altitude trekking population.

DETAILED DESCRIPTION:
The specific aim of this study is to evaluate if an inexpensive and disposable end-expiratory pressure device can prevent acute mountain sickness (AMS). AMS is a common disorder found in 25-75% of hikers and trekkers in N. America and Europe who expediently ascend high altitude (>8,000 ft). This environmental malady is insidious in onset and prevention is necessary not just to limit progression to severe or fatal disease, but also to limit physiologic deterioration in those who seek enjoyment or employment at high altitudes. One of the hallmarks of both healthy and sick individuals sleeping at high altitude is an oscillating pattern of respiration marked by periods of hyperventilation alternating with apnea or hypopnea. This distressing "periodic breathing" pattern leads to a feeling of suffocation, prevents restful sleep, and the hypoxic events may well worsen ensuing AMS. Prior studies have found positive end-expiratory pressure (PEEP) an effective non-pharmacologic method to prevent nocturnal desaturations and decreasing both AMS incidence and severity.

Traditionally, PEEP devices are cumbersome and expensive, and while showing promising efficacy, are limited by both cost and portability as a useful non-pharmacologic option for AMS prophylaxis. The SLEEP-AID methodology is designed to prospectively enroll participants, randomized in a double blind placebo-controlled fashion to either the intervention [Theravent (Ventus Medical) which is single use, inexpensive, and very small] or a visually identical "sham" placebo group, and gather physiologic data to accurately reflect sleep patterns of high altitude travelers and objective as well as subjective outcomes of the intervention. The benefit of this approach will be to provide definitive data in a large and diverse cross section of a real hiking population that is generalizable to the majority of tens of millions of hikers, climbers, and high altitude tourists in the United States, Europe, Asia, and South America.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* Lake Louise Score (LLS) of < 3
* Have not taken NSAIDs, acetazolamide, or corticosteroids in the prior week
* Have not traveled above 4200 m in the prior week.
* First night in Pheriche or Dingboche

Exclusion Criteria:

* Unable to read the consent form
* Taken NSAIDs, acetazolamide, or corticosteroids in the week prior to study enrollment.
* Hazardous medical conditions which precludes the ability to tolerate the experimental device.
* Pregnancy or suspected pregnancy.
* Participants who are younger than 18 years of age and more than 65.
* Travel to or above 4200m in the preceding week.
* Diagnosis of AMS upon enrollment (LLS ≥3 with symptoms of headache)
* Previously diagnosed obstructive sleep apnea
* Current symptoms of nasal congestion, rhinorrhea, sinusitis, upper respiratory infection, asthma, COPD exacerbation, pneumonia, bronchitis, or other disease of the respiratory tract.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Actual)
Dates: Start 2013-10; Primary Completion 2013-12 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant S Lipman, MD, Principal Investigator — Stanford University
Locations (1):
- Nepal, Pheriche & Dingboche, Khumbu, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lipman GS, Kanaan NC, Phillips C, Pomeranz D, Cain P, Fontes K, Higbee B, Meyer C, Shaheen M, Wentworth S, Walsh D. Study Looking at End Expiratory Pressure for Altitude Illness Decrease (SLEEP-AID). High Alt Med Biol. 2015 Jun;16(2):154-61. doi: 10.1089/ham.2014.1110. Epub 2015 May 7. PMID 25950723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Theravent | Control
Started | 115 | 104
Completed | 115 | 104
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Theravent | Control | Total
Number analyzed (Participants) | 115 | 104 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (6) | 37 (8) | 38 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 83 | 73 | 156
Region of Enrollment [Number; unit: participants]
  Nepal | 115 | 104 | 219

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Acute Mountain Sickness
Description: Acute mountain sickness will be measured by Lake Louise Criteria and diagnosed as LLC > or = to 3 with presence of a headache. Study participants will be followed approximately for 10 hours, from when they go to sleep until awakening the next morning.
Time Frame: Approximately 10 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Theravent
Number analyzed (Participants) | 104 | 115
Participants | 18 | 16

2. Secondary Outcome: Number of Nocturnal Desaturations
Description: Number of nocturnal desaturations will be measured by Watch-PAT200, a wristwatch type continuous sleep cycle and pulse oximetry analyzer. Study participants will be followed approximately for 10 hours, from when they go to sleep until awakening the next morning.
Time Frame: Approximately 10 hours
Measure: Mean (Standard Deviation); unit: Number of events
Arm/Group | Control | Theravent
Number analyzed (Participants) | 104 | 115
Number of events | 270 (226) | 214 (183)

3. Secondary Outcome: Acute Mountain Sickness Severity
Description: Severity of acute mountain sickness will be evaluated by the Lake Louise Criteria (0-15 point scale) with higher scores representing more severe symptoms. Study participants will be followed approximately for 10 hours, from when they go to sleep until awakening the next morning.
Time Frame: approximately 10 hours
Population: Severity
Measure: Median (Inter-Quartile Range); unit: unit on a scale
Arm/Group | Control | Theravent
Number analyzed (Participants) | 104 | 115
unit on a scale
  Headache severity | 0.46 [0 to 3] | 0.26 [0 to 3]
  Fatigue severity | 0.15 [0 to 2] | 0.20 [0 to 2]
  Dizziness severity | 0.15 [0 to 1] | 0.049 [0 to 1]
  Sleep severity | 1.11 [0 to 3] | 1.13 [0 to 3]
  Gastrointestinal symptoms severity | 0.11 [0 to 1] | 0.058 [0 to 1]

4. Secondary Outcome: Nocturnal Awakenings
Description: as for outcome 2
Time Frame: approximately 10 hours
Measure: Median (Inter-Quartile Range); unit: Number of events
Arm/Group | Control | Theravent
Number analyzed (Participants) | 104 | 115
Number of events | 11 [6 to 14] | 13 [7 to 18]

ADVERSE EVENTS:
Time Frame: 2 months (duration of study and intervention)
Arm/Group | Control | Theravent
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/115
Other Adverse Events (participants affected / at risk) | 0/104 | 0/115

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No